CLINICAL TRIAL: NCT03744507
Title: A Prospective Observational Study of Bone Mineral Density in Women With Uterine Fibroids or Endometriosis
Brief Title: Bone Mineral Density in Women With Uterine Fibroids or Endometriosis
Status: Completed | Type: Observational
Sponsor: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MVT-601-034; 2018-001367-22 (EudraCT Number)
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Uterine Fibroid; Endometriosis
Keywords: Uterine leiomyoma; Uterine fibroids; Heavy menstrual bleeding; Menorrhagia; Endometriosis
MeSH Terms: conditions — Leiomyoma; Endometriosis; Myofibroma; Menorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uterine Fibroids: Premenopausal women with uterine fibroids confirmed by an ultrasound.
- Endometriosis: Premenopausal women with endometriosis diagnosed or confirmed by surgical or direct visualization, or histopathology within 10 years of the Screening visit.

SUMMARY:
The purpose of this study is to characterize the longitudinal bone mineral density (BMD) in premenopausal women with uterine fibroids or endometriosis.

DETAILED DESCRIPTION:
This is a prospective observational study to characterize longitudinal BMD of premenopausal women with uterine fibroids or endometriosis over the 52-week observational period.

Approximately 660 participants will be recruited into two cohorts: (1) premenopausal women with uterine fibroids confirmed by an ultrasound (approximately 260 participants), and (2) premenopausal women with endometriosis diagnosed or confirmed by surgical or direct visualization, or histopathology within 10 years of the Screening visit (approximately 400 participants).

Since age is a strong risk factor for BMD change over time, participants in this observational study will be matched by age category (18 to 24, 25 to 34, 35 to 44, and ≥45 years old), with participants enrolled in the interventional studies of relugolix.

During the Screening/Baseline period, the participant should be assessed for eligibility, and baseline dual-energy X-ray absorptiometry (DXA) scan will be obtained. Bone densitometry (lumbar spine [L1-L4], total hip, and femoral neck) will be obtained and submitted for central reading at Baseline, Week 24, and Week 52.

Information related to health care utilization for uterine fibroids or endometriosis and concomitant medications will be collected at every visit and during the phone calls at Week 12 and Week 36.

Collection of adverse events in this study will be limited to protocol-specified procedure-related adverse events. Reports of pregnancy will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Is a premenopausal female 18 to 50 years old
2. By the participant's report, had two consecutive regular menstrual cycles immediately prior to enrollment in the study. Participants with hormonal intrauterine devices or on other hormonal contraception methods that disrupt cyclic bleeding are not required to have two consecutive regular menstrual cycles.
3. Has one of the following conditions:

   1. Diagnosis of uterine fibroids that is confirmed by an ultrasound within 5 years prior to screening.
   2. Diagnosis of endometriosis confirmed by surgical or direct visualization and/or histopathologic confirmation.
4. Has not and is not expected to undergo a surgical procedure with bilateral oophorectomy within the 12 months following enrollment.

   Exclusion Criteria:
5. Has a weight that exceeds the weight limit of the dual-energy X-ray absorptiometry scanner
6. Has a baseline BMD z-score < -2.0 at spine, total hip, or femoral neck
7. Has a history of or currently has osteoporosis, or other metabolic bone disease
8. Use within the past 3 months prior to Screening or anticipated use of systemic glucocorticoids
9. Is currently pregnant or lactating, or intends to become pregnant during the study period

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Women with endometriosis or with uterine fibroids
Sampling Method: Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage change in Bone Mineral Density (BMD) in lumbar spine (L1-L4). | from Baseline up to Week 52
  Assessed by dual-energy X-ray absorptiometry (DXA) scan.
Percentage change in BMD in the femoral neck and total hip. | from Baseline up to Week 52
  Assessed by DXA scan.
Absolute change in BMD in the lumbar spine (L1-L4), femoral neck and total hip. | from Baseline up to Week 52
  Assessed by dual-energy X-ray absorptiometry (DXA) scan.

SECONDARY OUTCOMES:
Healthcare utilization for uterine fibroids or endometriosis | over 52 weeks
  Assessed through participants self-reporting (may be aided by review of participant medical records). Healthcare utilization includes visits to gynecologists or other primary care providers, visits to urgent care, visits to emergency department, hospitalizations, procedures (diagnostic or surgical) or changes to medication concomitant related to uterine fibroids or endometriosis.
Frequency of concomitant medication use. | over 52 weeks
  Assessed through participants self-reporting.
Change from Baseline on the European Quality of Life-5 Dimensions 5 Levels (EQ-5D-5L). | from Baseline up to Week 52
  Assessed using participants responses on the EQ-5D-5L questionnaire. The EQ-5D-5L is a standardized measure of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses (from 1= no problem to 5= extreme problems).

CONTACTS AND LOCATIONS:
Locations (55):
- United States (35):
  - Mobile, Mobile, Alabama
  - Mesa, Mesa, Arizona
  - Huntington Beach, Huntington Beach, California
  - Palos Verdes Estates, Palos Verdes Estates, California
  - Denver, Denver, Colorado
  - United States, Colorado, Denver, Colorado
  - Aventura, Aventura, Florida
  - Jupiter, Jupiter, Florida
  - Loxahatchee, Loxahatchee Groves, Florida
  - Margate, Margate, Florida
  - Miami, Miami, Florida
  - Orange City, Orange City, Florida
  - Orlando, Orlando, Florida
  - Port St. Lucie, Port Saint Lucie, Florida
  - Sarasota, Sarasota, Florida
  - West Palm Beach, West Palm Beach, Florida
  - Atlanta, Atlanta, Georgia
  - Decatur, Decatur, Georgia
  - Norcross, Norcross, Georgia
  - Oak Brook, Oak Brook, Illinois
  - Towson, Towson, Maryland
  - Canton, Canton, Michigan
  - Durham, Durham, North Carolina
  - Raleigh, Raleigh, North Carolina
  - Winston-Salem, Winston-Salem, North Carolina
  - Columbus, Columbus, Ohio
  - Chattanooga, Chattanooga, Tennessee
  - Memphis, Memphis, Tennessee
  - Beaumont, Beaumont, Texas
  - Fort Worth, Fort Worth, Texas
  - Houston, Houston, Texas
  - San Antonio, San Antonio, Texas
  - Sugar Land, Sugar Land, Texas
  - Webster, Webster, Texas
  - Virginia Beach, Virginia Beach, Virginia
- Australia (4):
  - Blacktown, Blacktown, New South Wales
  - Kanwal, Kanwal, New South Wales
  - Sherwood, Sherwood, Queensland
  - Nedlands, Nedlands, Western Australia
- Santiago, Santiago, Chile
- Czechia (3):
  - Pisek, Písek, Jihočeský kraj
  - Praha 10, Prague, Prague
  - Olomouc, Olomouc, Severomoravsky KRAJ
- Georgia (2):
  - Tbilisi, Tbilisi, Borjomi
  - Tbilisi, Tbilisi
- Hungary (4):
  - Gyula, Gyula, Bekes County
  - Kecskemet, Kecskemét, Bács-Kiskun county
  - Szeged, Szeged, Csongrád megye
  - Debrecen, Debrecen, Hajdú-Bihar
- Poland (6):
  - Skorzewo, Skórzewo, Greater Poland Voivodeship
  - Lublin, Lublin, Lublin Voivodeship
  - Warszawa, Warsaw, Masovian Voivodeship
  - Biaystok, Bialystok, Podlaskie Voivodeship
  - Katowice, Katowice, Silesian Voivodeship
  - Szczecin, Szczecin, West Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: No